CLINICAL TRIAL: NCT07391631
Title: The Relationship Between Preoperative and Postoperative Fasting Durations and Postoperative Delirium
Brief Title: Preoperative and Postoperative Fasting and Delirium
Acronym: FAST-POD
Status: Not yet recruiting | Type: Observational
Sponsor: Akdeniz University (Other)
Collaborators: Turkish Society of Anesthesiology and Reanimation (Other)
Responsible Party: Principal Investigator, Emel Gunduz, Associate Professor of Anesthesiology, Akdeniz University, Antalya, Turkey, Akdeniz University
Other Study IDs: TARD_FASTING_POD_01
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Delirium Perioperative Fasting
Keywords: Postoperative Delirium; Preoperative Fasting; Postoperative Fasting; Surgical Patients; Observational Study; Multicenter Study
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative delirium is a common and serious complication after surgery, especially in older patients, and is associated with prolonged hospital stay and worse recovery. Fasting before and after surgery is a routine part of perioperative care; however, prolonged fasting may negatively affect recovery and brain function.

This prospective, observational, multicenter study aims to evaluate the relationship between preoperative and postoperative fasting durations and the development of postoperative delirium in adult patients undergoing elective or emergency surgery under general or regional anesthesia.

Fasting times before and after surgery will be recorded. Patients will be assessed for postoperative delirium during the first three postoperative days using validated screening tools. No additional interventions will be applied, and all patients will receive standard perioperative care.

The results of this study may help identify whether prolonged fasting is associated with a higher risk of postoperative delirium and may contribute to improving perioperative fasting practices and patient safety.

DETAILED DESCRIPTION:
This is a prospective, observational, multicenter study designed to investigate the association between preoperative and postoperative fasting durations and the occurrence of postoperative delirium in adult surgical patients.

Adult patients (≥18 years) undergoing elective or emergency surgery under general or regional anesthesia will be included. Patients with pre-existing delirium, advanced dementia, postoperative intensive care unit admission, or inability to complete delirium assessments will be excluded.

Preoperative fasting duration will be defined as the time from the last oral intake to the induction of anesthesia. Postoperative fasting duration will be defined as the time from the end of surgery to the first oral intake. Fasting durations will be recorded for each participant.

Postoperative delirium will be assessed using validated screening tools (Confusion Assessment Method or Nursing Delirium Screening Scale) twice daily during the first three postoperative days. Routine perioperative management will not be altered for study purposes, and no study-specific interventions will be applied.

Demographic data, comorbidities, type of surgery, and perioperative clinical parameters will be collected as part of standard care. The primary objective is to evaluate the relationship between fasting durations and postoperative delirium. Secondary analyses will explore factors associated with delirium development.

ELIGIBILITY:
Inclusion Criteria:Adults aged 18 years or older

Patients undergoing elective or emergency surgery under general or regional anesthesia

Ability to communicate and cooperate with postoperative delirium assessments

Expected postoperative hospital stay of at least 72 hours

Provision of written informed consent

-

Exclusion Criteria:Presence of preoperative delirium (positive CAM or Nu-DESC ≥2)

Advanced dementia or severe cognitive impairment

Planned postoperative intensive care unit admission

Active alcohol or benzodiazepine withdrawal

Inability to complete delirium assessments due to severe hearing, vision, or speech impairment

Lack of postoperative follow-up availability

Planned cardiac surgery

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older who undergo elective or emergency surgical procedures under general or regional anesthesia. Participants are hospitalized for postoperative follow-up and are assessed prospectively for fasting durations and postoperative delirium as part of routine perioperative care.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | During the first 3 postoperative days
  Postoperative delirium will be assessed using validated screening tools (Confusion Assessment Method or Nursing Delirium Screening Scale) during the first three postoperative days.

SECONDARY OUTCOMES:
Duration of postoperative delirium | During the first 3 postoperative days
  The duration of postoperative delirium will be recorded based on daily delirium assessments during the first three postoperative days.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study is observational and data are collected for predefined research purposes in accordance with local ethical approval and data protection regulations.